CLINICAL TRIAL: NCT04047134
Title: Neuroimaging Biomarkers Toward an Optimized and Personalized Action Observation Treatment in Chronic Stroke Patients: New Strategies to Maximize the Efficacy of Upper Limb Functional Rehabilitation.
Brief Title: Neuroimaging Biomarkers Toward a Personalized Upper Limb Action Observation Treatment in Chronic Stroke Patients
Acronym: BE-TOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Casa di Cura del Policlinico di Milano (Unknown)
Responsible Party: Principal Investigator, Francesco Infarinato, Responsible of Rehab-bioengeneering lab., IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05/2018; GR-2016 - 02361678 (Other Grant/Funding Number: Italian Ministery of Health)
Record Dates: First submitted 2019-07-31; First posted 2019-08-06 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Chronic Stroke
Keywords: Prevention and treatment of movement; Motor Function; Action Observation Therapy; Mirror Neuron System; Upper Limb Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (EG) (Experimental): The Experimental Group (EG) will observe and execute/repeat Activities of Daily Living (ADL) actions.
  Interventions: Other: Action Observation Treatrment
- Control Group (CG) (Active Comparator): The COntrol Group (CG) will observe landscapes and perform the same actions observed by their peers but after verbal instructions.
  Interventions: Other: Observation of videos with Non Motor contents

INTERVENTIONS:
Other: Action Observation Treatrment — Participants will be asked to carefully observe the videos showing different daily actions. Each action will consist of 3 to 4 constituent motor acts. Each motor act will be presented for 3 minutes, totally lasting 12 min/video. At the end of each motor act presentation, participants will be asked to execute with the affected hand the observed motor sequence for 2 minutes (20 minutes/session). 10 daily actions will be recorded. Each video will be presented to participants twice a day, in order to complexity as judged by the experimenter. Only 1 typology of motor task per day for each condition, starting from the easiest and ending with the most complex action throughout 15 sessions spread on 5 weeks (3 sessions/week). Tasks will be based on some relevant activities of daily living belonging to at least one between feeding, self-care or external actions category on the affected side. Each session will last about 15 minutes and will be repeated twice a day, at least 60 minutes apart.
  Other Names: AOT
  Arms: Experimental Group (EG)
Other: Observation of videos with Non Motor contents — Participants will be asked to observe video clips with no specific motor content. Videos will concern scientific, geographical and historical issues. As for cases, video clips will be divided into three to four parts. At the end of each part, controls will execute the same actions as cases, in the same order. In this way cases and controls will undergo the same amount of motor practice and receive the same amount of visual stimulation, the only difference being the content of visual stimuli.
  Other Names: NMO
  Arms: Control Group (CG)

SUMMARY:
Much recent interest was raised by the use of Action Observation Treatment (AOT) in stroke patients rehabilitation. AOT, well-grounded in neurophysiology, is an updated approach, based on mirror neuron system (MNS) used to rebuild motor function despite injuries by engaging the brain regions active during action execution in individuals with limited mobility. This project aims at identifying, for the first time in Italy, neurophysiological electroencephalographic (EEG) biomarkers able to predict rehabilitation outcomes and providing an innovative optimized AOT rehabilitation protocol for chronic Stroke outpatients. EEG will be recorded to identify the most effective stimuli, quantify changes/recovery, profile patients.

Moreover, an innovative AOT home-based program will be implemented. The translational research results will ensure advances in the optimization and personalization of the rehabilitative process thus contributing to improve the quality of life of chronic stroke patients.

Stroke is a leading cause of death and one of the greatest causes of long-term disability that interferes with a good quality of life. Nowadays the rehabilitation interventions are the major component of patient's care to achieve functional outcome. In the last few years, in order to improve Activity of Daily Living (ADL), new noninvasive strategies have emerged as rehabilitative treatments rather than traditional physical therapies. The Action Observation Treatment (AOT), supported by results collected through randomized controlled trials, is one of these. This new rehabilitation approach is based on the properties of the Mirror Neuron System (MNS; 11-13). The extensive research of the last 20 years on the human MNS (hMNS) showed its importance not only in action recognition but also in motor intentions and other social cognitive functions. Lastly, because recruited also in damage brain (18,19), the MNS is demonstrated to provide satisfactory rehabilitative outcomes. The AOT takes advantage of the opportunity to restore functions despite the patient's impairment and it seems to be a valid example of translational medicine from basic neuroscience to rehabilitation. To date, neurophysiological outcomes were never used for translational purposes aimed to the optimization of the therapy and no evidence, in Italy, related to the effectiveness of the home-based program were proposed.

DETAILED DESCRIPTION:
This study protocol provides 3 experimental designs to satisfy 3 different specific aims as follows.

Experimental design aim 1:

To assess which kind of ADL visual stimuli will be most effective inducing motor excitability during action observation, EEG recording will be performed. 20 Stroke patients (10 with right lesion and 10 left one) will be recruited and video of feeding, self care and external actions showed. The EEG biomarkers will be identify. A comparison on EEG rhythm and biomarkers between the two groups and the ADL categories observed will be investigated. The most effective category will be subsequently selected for the Randomized Controlled Trial (RCT).

Experimental design aim 2:

This is an RCT study aimed to deeply investigate if EEG biomarkers are predictive of effectiveness of AOT on 40 Chronic Stroke outpatients in order to confirm the translational power of the optimized treatment. The subjects accurately enrolled for hospital program, will be randomly assigned to the Experimental Group (EG) or to the Control one (CG). The EG will observe and execute ADL actions, the CG will observe landscapes and perform the same actions observed by the others one but after verbal instructions. For each condition the patient will be presented with only 1 typology of motor task per day, starting from the easiest and ending with the most complex action throughout 15 sessions spread on 5 weeks (3 sessions/week). Tasks will be based on some relevant activities of daily living belonging to at least one between feeding, self-care or external actions category on the affected side. Each session will last about 15 minutes and will be repeated twice a day, at least 60 minutes apart. Before, after and in the middle of the treatment sessions all patients will be clinically, neurophysiologically (EEG and EMG) and behaviorally (Kinematics) assessed to verify neural plasticity and motor recovery.

The follow-up at 2 months later will be carried out to assess retention of effects.

Experimental design aim 3:

The health policy to develop appropriate home-based rehabilitation programs for chronic stroke patients (24,25) could induce to explore whether AOT can meet the necessary translational requirements also for this type of care. A New group of 20 chronic stroke patients will be recruited and randomly assigned to the EG OR CG to follow the optimized AOT rehabilitation programs.

After appropriate training of patients and caregivers, the use of tablets will let the home-based treatment. The investigators will define a low-cost highly accessible system based on tablet consumer technology for facilitating the AOT. In particular a tablet will be proposed with a web-based program that will be used to train the patients and receive a feedback of their progress.

The whole treatment period will last 6 weeks. The focus of this evaluation will be on the feasibility of the home-based treatment and the usability of the platform as well as the subjects satisfaction with the services. A preliminary estimate of the recovery and overall improvement of functional performances of participants will also be provided with respect to clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* chronic stroke (never experienced AOT);
* first-ever unilateral stroke due to ischemia provoking a clinically evident upper limb/hand deficit;
* diagnosis verified by brain imaging (MRI);
* cognitive function sufficient to understand the experimental instructions
* Chedoke-McMaster stroke Assessment Scale score greater than 1;
* informed written consent to participate in the study.

Exclusion Criteria:

* bilateral impairment,
* severe sensory deficits in the paretic upper limb,
* cognitive impairment or behavioral dysfunction,
* refusal or inability to provide informed consent and
* other current severe medical problems.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer (FM) Test | At baseline-day 0 (T0), the middle of the treatment-day 15 (T1), at the end treatment-day 30 (T2), and at the follow up visit-day 90 (2 months both for the hospital-based and for the home based program) (T3)
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment. The scale is comprised of five domains and there are 155 items in total:
  * Motor functioning (the score ranges from 0 (hemiplegia) to 100 points (normal motor performance). Divided into 66 points for upper extremity and 34 points for the lower extremity.
  * Sensory functioning (from 0 to 24 points)
  * Balance (from 0 to 14)
  * Joint range of motion (from 0 to 44)
  * Joint pain (from 0 to 44 ) Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully. The total possible scale score is 226.

SECONDARY OUTCOMES:
Change in Frenchay Arm Test (FAT) | At baseline-day 0 (T0), the middle of the treatment-day 15 (T1), at the end treatment-day 30 (T2), and at the follow up visit-day 90 (2 months both for the hospital-based and for the home based program) (T3)
  The Frenchay Arm Test (FAT) is a measure of upper extremity proximal motor control and dexterity during ADL performance in patients with impairments resulting from neurological conditions. The FAT is an upper extremity specific measure of activity limitation.

OTHER OUTCOMES:
Change in Box and Block Test (BBT) | At baseline-day 0 (T0), the middle of the treatment-day 15 (T1), at the end treatment-day 30 (T2), and at the follow up visit-day 90 (2 months both for the hospital-based and for the home based program) (T3)
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. It is a quick, simple and inexpensive test. It can be used with a wide range of populations, including clients with stroke.
Change in Modified Ashworth Scale (MSA) | At baseline-day 0 (T0), the middle of the treatment-day 15 (T1), at the end treatment-day 30 (T2), and at the follow up visit-day 90 (2 months both for the hospital-based and for the home based program) (T3)
  The Modified Ashworth scale (MAS) measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity.[1] Scoring (taken from Bohannon and Smith, 1987):
  0: No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the Range Of Motion (ROM)
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
Change in Modified Bartel Index (mBI) | At baseline-day 0 (T0), the middle of the treatment-day 15 (T1), at the end treatment-day 30 (T2), and at the follow up visit-day 90 (2 months both for the hospital-based and for the home based program) (T3)
  The Modified Bartel Index (mBI) is an ordinal scale used to measure performance in activities of daily living (ADL). Each performance item is rated on this scale with a given number of points assigned to each level or ranking. It uses ten variables describing ADL and mobility. A higher number is associated with a greater likelihood of being able to live at home with a degree of independence following discharge from hospital.
Change in Chedoke-McMaster Stroke Assessment scale | At baseline-day 0 (T0), the middle of the treatment-day 15 (T1), at the end treatment-day 30 (T2), and at the follow up visit-day 90 (2 months both for the hospital-based and for the home based program) (T3)
  The Chedoke-McMaster Stroke Assessment measures physical impairment and disability in people with stroke and other neurological impairment. The measure consists of an Impairment Inventory and an Activity Inventory (Moreland, Gowland, Van Hullenaar, & Huijbregts, 1993). The first inventory aims to determine the presence and severity of common physical impairments, to classify or stratify patients when planning, selecting interventions and evaluating their effectiveness and to predict outcomes. The second inventory measures changes in physical function (Gowland, Stratford, Ward, Moreland, Torresin, Van Hullenar, Sanford, Barreca, Vanspall, & Plews, 1993).
  No helper needed 7 Complete Independence (Timely, Safely) 6 Modified Independence 5 Supervision A helper needed 4 Minimal Assist (Client = 75%) 3 Moderate Assist (Client = 50%) Complete Dependence 2 Maximal Assist (Client = 25%)
  1 Total Assist (Client = 0%)
Change in Mini-Mental state examination (MMSE) | At baseline-day 0 (T0), at the end treatment-day 30 (T2) and at the follow up visit-day 90 (2 months both for the hospital-based and for the home based program) (T3)
  Il Mini-Mental State Examination (MMSE) (Folstein et al., 1975), is a neuropsychological test for the assessment of intellectual efficiency disorders and the presence of cognitive deterioration.
  The total score is between a minimum of 0 and a maximum of 30 points, where a score of 30 represents the best cognitive condition, and 0 the worst.
  The Mini-Mental state examination (MMSE) is often used as a screening tool in the investigation of subjects with dementia, and with neuropsychological syndromes of different nature.
Change in ElectroEncephaloGraphy (EEG) | At baseline-day 0 (T0), at the end treatment-day 30 (T2) and at the follow up visit-day 90 (2 months both for the hospital-based and for the home based program) (T3)
  Electroencephalography (EEG) is an electrophysiological monitoring method to record electrical activity of the brain. It is noninvasive, with the electrodes placed over the scalp. Each conscious and unconscious mental function is the result of the electrical communication among the human brain neurons. It is not possible to record in a no-invasive way the electrical activity related to each neuron, however the EEG technique is able to measure the voltage fluctuations over the scalp caused by the concomitant electrical activity of a neurons population. Such voltage fluctuations could be characterized in terms of spectral content (EEG rhythms or bands) or of time-domain characteristics (Evoked Potentials and Event-Related Potentials). Alph (8-13 Htz), Beta (14-30 Htz) and Mu (8-13 Htz) bandwidth will be registered. The last band will be analysed specifically to investigate the motor areas and mirror neuron system's activity.
Change in surface ElectroMioGraphy (sEMG) - arm and shoulder muscles | At baseline-day 0 (T0), at the end treatment-day 30 (T2) and at the follow up visit-day 90 (2 months both for the hospital-based and for the home based program) (T3)
  Surface electromyography (sEMG) is a non-invasive procedure involving the detection, recording and interpretation of the electric activity of groups of muscles at rest (i.e., static) and during activity (i.e., dynamic). The procedure is performed using a single or an array of electrodes placed on the skin surface over the muscles to be tested. Recording can also be made using a hand-held device, which is applied to the skin surface at different sites. Electrical activity is assessed by computer analysis of the frequency spectrum, amplitude, or root mean square of the electrical action potential.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Infarinato, Phd, Study Chair — IRCSS San Raffaele Pisana
Locations (2):
- Italy (2):
  - Casa di Cura del Policlinico di Milano, Milan, MI
  - IRCCS San Raffaele Pisana, Rome, RM

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gosman-Hedstrom G, Claesson L, Blomstrand C. Consequences of severity at stroke onset for health-related quality of life (HRQL) and informal care: a 1-year follow-up in elderly stroke survivors. Arch Gerontol Geriatr. 2008 Jul-Aug;47(1):79-91. doi: 10.1016/j.archger.2007.07.006. Epub 2007 Sep 14. PMID 17868935
- [Background] Laver KE, George S, Thomas S, Deutsch JE, Crotty M. Virtual reality for stroke rehabilitation. Cochrane Database Syst Rev. 2011 Sep 7;(9):CD008349. doi: 10.1002/14651858.CD008349.pub2. PMID 21901720
- [Background] Pollock A, Farmer SE, Brady MC, Langhorne P, Mead GE, Mehrholz J, van Wijck F. Interventions for improving upper limb function after stroke. Cochrane Database Syst Rev. 2014 Nov 12;2014(11):CD010820. doi: 10.1002/14651858.CD010820.pub2. PMID 25387001
- [Background] Michielsen ME, Selles RW, van der Geest JN, Eckhardt M, Yavuzer G, Stam HJ, Smits M, Ribbers GM, Bussmann JB. Motor recovery and cortical reorganization after mirror therapy in chronic stroke patients: a phase II randomized controlled trial. Neurorehabil Neural Repair. 2011 Mar-Apr;25(3):223-33. doi: 10.1177/1545968310385127. Epub 2010 Nov 4. PMID 21051765
- [Background] Ertelt D, Small S, Solodkin A, Dettmers C, McNamara A, Binkofski F, Buccino G. Action observation has a positive impact on rehabilitation of motor deficits after stroke. Neuroimage. 2007;36 Suppl 2:T164-73. doi: 10.1016/j.neuroimage.2007.03.043. Epub 2007 Mar 31. PMID 17499164
- [Background] Franceschini M, Agosti M, Cantagallo A, Sale P, Mancuso M, Buccino G. Mirror neurons: action observation treatment as a tool in stroke rehabilitation. Eur J Phys Rehabil Med. 2010 Dec;46(4):517-23. Epub 2010 Apr 23. PMID 20414184
- [Background] Franceschini M, Ceravolo MG, Agosti M, Cavallini P, Bonassi S, Dall'Armi V, Massucci M, Schifini F, Sale P. Clinical relevance of action observation in upper-limb stroke rehabilitation: a possible role in recovery of functional dexterity. A randomized clinical trial. Neurorehabil Neural Repair. 2012 Jun;26(5):456-62. doi: 10.1177/1545968311427406. Epub 2012 Jan 10. PMID 22235059
- [Background] Buccino G, Arisi D, Gough P, Aprile D, Ferri C, Serotti L, Tiberti A, Fazzi E. Improving upper limb motor functions through action observation treatment: a pilot study in children with cerebral palsy. Dev Med Child Neurol. 2012 Sep;54(9):822-8. doi: 10.1111/j.1469-8749.2012.04334.x. Epub 2012 Jul 6. PMID 22765352
- [Background] Brunner IC, Skouen JS, Ersland L, Gruner R. Plasticity and response to action observation: a longitudinal FMRI study of potential mirror neurons in patients with subacute stroke. Neurorehabil Neural Repair. 2014 Nov-Dec;28(9):874-84. doi: 10.1177/1545968314527350. Epub 2014 Mar 18. PMID 24642381
- [Background] Gallese V, Fadiga L, Fogassi L, Rizzolatti G. Action recognition in the premotor cortex. Brain. 1996 Apr;119 ( Pt 2):593-609. doi: 10.1093/brain/119.2.593. PMID 8800951
- [Background] Fogassi L, Ferrari PF, Gesierich B, Rozzi S, Chersi F, Rizzolatti G. Parietal lobe: from action organization to intention understanding. Science. 2005 Apr 29;308(5722):662-7. doi: 10.1126/science.1106138. PMID 15860620
- [Background] Bonini L, Rozzi S, Serventi FU, Simone L, Ferrari PF, Fogassi L. Ventral premotor and inferior parietal cortices make distinct contribution to action organization and intention understanding. Cereb Cortex. 2010 Jun;20(6):1372-85. doi: 10.1093/cercor/bhp200. Epub 2009 Oct 5. PMID 19805419
- [Background] Campione GC, Gentilucci M. Is the observation of the human kinematics sufficient to activate automatic imitation of transitive actions? Behav Brain Res. 2011 Nov 20;225(1):201-8. doi: 10.1016/j.bbr.2011.07.025. Epub 2011 Jul 23. PMID 21802449
- [Background] Rizzolatti G, Sinigaglia C. The functional role of the parieto-frontal mirror circuit: interpretations and misinterpretations. Nat Rev Neurosci. 2010 Apr;11(4):264-74. doi: 10.1038/nrn2805. Epub 2010 Mar 10. PMID 20216547
- [Background] Rizzolatti G, Cattaneo L, Fabbri-Destro M, Rozzi S. Cortical mechanisms underlying the organization of goal-directed actions and mirror neuron-based action understanding. Physiol Rev. 2014 Apr;94(2):655-706. doi: 10.1152/physrev.00009.2013. PMID 24692357
- [Background] Bonini L, Ferrari PF, Fogassi L. Neurophysiological bases underlying the organization of intentional actions and the understanding of others' intention. Conscious Cogn. 2013 Sep;22(3):1095-104. doi: 10.1016/j.concog.2013.03.001. Epub 2013 Mar 30. PMID 23545395
- [Background] Frenkel-Toledo S, Bentin S, Perry A, Liebermann DG, Soroker N. Mirror-neuron system recruitment by action observation: effects of focal brain damage on mu suppression. Neuroimage. 2014 Feb 15;87:127-37. doi: 10.1016/j.neuroimage.2013.10.019. Epub 2013 Oct 18. PMID 24140938
- [Background] Garrison KA, Aziz-Zadeh L, Wong SW, Liew SL, Winstein CJ. Modulating the motor system by action observation after stroke. Stroke. 2013 Aug;44(8):2247-53. doi: 10.1161/STROKEAHA.113.001105. Epub 2013 Jun 6. PMID 23743974
- [Background] Kuk EJ, Kim JM, Oh DW, Hwang HJ. Effects of action observation therapy on hand dexterity and EEG-based cortical activation patterns in patients with post-stroke hemiparesis. Top Stroke Rehabil. 2016 Oct;23(5):318-25. doi: 10.1080/10749357.2016.1157972. Epub 2016 Mar 31. PMID 27077994
- [Background] Buccino G. Action observation treatment: a novel tool in neurorehabilitation. Philos Trans R Soc Lond B Biol Sci. 2014 Apr 28;369(1644):20130185. doi: 10.1098/rstb.2013.0185. Print 2014. PMID 24778380
- [Background] Sale P, Franceschini M. Action observation and mirror neuron network: a tool for motor stroke rehabilitation. Eur J Phys Rehabil Med. 2012 Jun;48(2):313-8. Epub 2012 Apr 20. PMID 22522432
- [Background] Babiloni C, Del Percio C, Rossini PM, Marzano N, Iacoboni M, Infarinato F, Lizio R, Piazza M, Pirritano M, Berlutti G, Cibelli G, Eusebi F. Judgment of actions in experts: a high-resolution EEG study in elite athletes. Neuroimage. 2009 Apr 1;45(2):512-21. doi: 10.1016/j.neuroimage.2008.11.035. Epub 2008 Dec 10. PMID 19111623
- [Background] Laver KE, Schoene D, Crotty M, George S, Lannin NA, Sherrington C. Telerehabilitation services for stroke. Cochrane Database Syst Rev. 2013 Dec 16;2013(12):CD010255. doi: 10.1002/14651858.CD010255.pub2. PMID 24338496
- [Background] Chumbler NR, Quigley P, Li X, Morey M, Rose D, Sanford J, Griffiths P, Hoenig H. Effects of telerehabilitation on physical function and disability for stroke patients: a randomized, controlled trial. Stroke. 2012 Aug;43(8):2168-74. doi: 10.1161/STROKEAHA.111.646943. Epub 2012 May 24. PMID 22627983
- [Background] Li L, Wang J, Xu G, Li M, Xie J. The Study of Object-Oriented Motor Imagery Based on EEG Suppression. PLoS One. 2015 Dec 7;10(12):e0144256. doi: 10.1371/journal.pone.0144256. eCollection 2015. PMID 26641241
- [Background] Simis M, Doruk D, Imamura M, Anghinah R, Morales-Quezada L, Fregni F, Battistella LR. Neurophysiologic predictors of motor function in stroke. Restor Neurol Neurosci. 2016;34(1):45-54. doi: 10.3233/RNN-150550. PMID 26518670
- [Background] Kim J, Kim S. The effects of visual stimuli on EEG mu rhythms in healthy adults. J Phys Ther Sci. 2016 Jun;28(6):1748-52. doi: 10.1589/jpts.28.1748. Epub 2016 Jun 28. PMID 27390408
- [Background] Caimmi M, Visani E, Digiacomo F, Scano A, Chiavenna A, Gramigna C, Molinari Tosatti L, Franceschetti S, Molteni F, Panzica F. Predicting Functional Recovery in Chronic Stroke Rehabilitation Using Event-Related Desynchronization-Synchronization during Robot-Assisted Movement. Biomed Res Int. 2016;2016:7051340. doi: 10.1155/2016/7051340. Epub 2016 Jan 17. PMID 27057546
- [Derived] Tropea P, Infarinato F, Sterpi I, Ottaviani M, Antoniotti P, Romano P, Picardi M, Goffredo M, Re R, Pournajaf S, Seregni A, Caronni A, Franceschini M, Corbo M. Action Observation Treatment for Upper Limb Rehabilitation in Patients With Stroke: Protocol for a Multicenter Randomized Controlled Trial. JMIR Res Protoc. 2023 Apr 20;12:e42094. doi: 10.2196/42094. PMID 37079364
- [Derived] Franceschini M, Ottaviani M, Romano P, Goffredo M, Pournajaf S, Lofrumento M, Proietti S, Sterpi I, Tricomi E, Tropea P, Corbo M, Fadiga L, Infarinato F. The Reaching Phase of Feeding and Self-Care Actions Optimizes Action Observation Effects in Chronic Stroke Subjects. Neurorehabil Neural Repair. 2022 Sep;36(9):574-586. doi: 10.1177/15459683221110884. Epub 2022 Aug 24. PMID 36000699
- [Derived] Borges LR, Fernandes AB, Oliveira Dos Passos J, Rego IAO, Campos TF. Action observation for upper limb rehabilitation after stroke. Cochrane Database Syst Rev. 2022 Aug 5;8(8):CD011887. doi: 10.1002/14651858.CD011887.pub3. PMID 35930301